CLINICAL TRIAL: NCT00294801
Title: Effect of Flex-a-New on Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: flex-a-new
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Osteoarthritis
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Dietary Supplements

INTERVENTIONS:
Drug: flex-a-new (food supplement)

SUMMARY:
comparative trial of placebo versus flex-a-new (a food supplement) containing glucosamine an chondroitin sulfate for the symptom modification is knee osteoarthritis

DETAILED DESCRIPTION:
comparative trial of placebo versus flex-a-new (a food supplement) containing glucosamine an chondroitin sulfate for the symptom modification is knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

knee osteoarthritis grade 1 to 3 -

Exclusion Criteria:

ischemic heart disease with CHF -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-01; Study Completion 2007-12

PRIMARY OUTCOMES:
KOOS

SECONDARY OUTCOMES:
VAS KSS

CONTACTS AND LOCATIONS:
Overall Officials: dror robinson, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikwa, Israel